CLINICAL TRIAL: NCT02010996
Title: Preventing Seroma Formation After Stripping Saphenous Vein in Coronary Bypass - a Randomized Control Clinical Trial
Brief Title: Preventing Seroma Formation After Stripping Saphenous Vein in Coronary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Bi-Hongda, physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSF20131201
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Bypass Graft Stenosis of Autologous Vein
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vacuum assisted closure (Experimental): Vacuum assisted closure (also called vacuum therapy, vacuum sealing or topical negative pressure therapy) is a sophisticated development of a standard surgical procedure, the use of vacuum assisted drainage to remove blood or serous fluid from a wound or operation site.
  Interventions: Procedure: vacuum assisted closure
- Axillary dissection (Active Comparator): Axillary dissection is a surgical procedure that incises (opens) the armpit (axilla or axillary) to identify, examine, or remove lymph nodes (small glands, part of the lymphatic system, which filters cellular fluids).
  Interventions: Procedure: Axillary dissection

INTERVENTIONS:
Procedure: vacuum assisted closure — Vacuum assisted closure (also called vacuum therapy, vacuum sealing or topical negative pressure therapy) is a sophisticated development of a standard surgical procedure, the use of vacuum assisted drainage to remove blood or serous fluid from a wound or operation site.
  Arms: Vacuum assisted closure
Procedure: Axillary dissection — Axillary dissection is a surgical procedure that incises (opens) the armpit (axilla or axillary) to identify, examine, or remove lymph nodes (small glands, part of the lymphatic system, which filters cellular fluids).
  Arms: Axillary dissection

SUMMARY:
The great saphenous vein is the most commonly used material in coronary vascular bridging operation. Coronary bypass operation to obtain the great saphenous vein is mainly through the incision open groin to ankle. This operation may damage the lymphatic, cause lymph circumfluence obstacle, cause fat liquefaction, scar formation, wound dehiscence, around hematoma and other a series of symptoms.Based on some studies and our experience that vacuum assisted closure （VAC）is effective in complex wound failures following Stripping saphenous vein, we use VAC to prevent seroma formation after Stripping saphenous vein in Coronary bypass. This study is aimed to evaluate the efficacy and economics benefits of early VAC application on postoperative complications and wound healing after Stripping saphenous vein in Coronary bypass in comparison to conventional suction drain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Coronary heart disease patients to transplant more than 2 vascular bridge
* The thigh groin following from the saphenous vein

Exclusion Criteria:

* Subjects does not agree to participate in clinical trials
* Subjects had a injury, operation history of Thigh
* Subjects having ever received chemotherapy before the surgery
* Subjects with known hypersensitivity to components of the surgical sticky membrane

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: hongda bi, Ph.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu Y, Song Z, Xu Z, Ye X, Xue C, Li J, Bi H. Bilayered negative-pressure wound therapy preventing leg incision morbidity in coronary artery bypass graft patients: A randomized controlled trial. Medicine (Baltimore). 2017 Jan;96(3):e5925. doi: 10.1097/MD.0000000000005925. PMID 28099357

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vacuum Assisted Closure | Axillary Dissection
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vacuum Assisted Closure | Axillary Dissection | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.2) | 55.4 (12.4) | 56.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 25 | 23 | 48
diabetes [Number; unit: participants]
  yes | 17 | 16 | 33
  no | 19 | 20 | 39
carotid artery stenosis [Number; unit: participants]
  yes | 5 | 4 | 9
  no | 31 | 32 | 63
smoking [Number; unit: participants]
  yes | 20 | 21 | 41
  no | 16 | 15 | 31
obesity [Number; unit: participants]
  yes | 8 | 6 | 14
  no | 28 | 30 | 58
glucocorticoid [Number; unit: participants]
  yes | 1 | 0 | 1
  no | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Early Complications of Vascular Zone
Time Frame: 2 weeks
Measure: Number; unit: participants
Groups:
- Vacuum Assisted Closure(Thigh): Vacuum assisted closure (also called vacuum therapy, vacuum sealing or topical negative pressure therapy) is a sophisticated development of a standard surgical procedure, the use of vacuum assisted drainage to remove blood or serous fluid from a wound or operation site.
  vacuum assisted closure: Vacuum assisted closure (also called vacuum therapy, vacuum sealing or topical negative pressure therapy) is a sophisticated development of a standard surgical procedure, the use of vacuum assisted drainage to remove blood or serous fluid from a wound or operation site.
- Axillary Dissection(Thigh): Axillary dissection is a surgical procedure that incises (opens) the armpit (axilla or axillary) to identify, examine, or remove lymph nodes (small glands, part of the lymphatic system, which filters cellular fluids).
  Axillary dissection: Axillary dissection is a surgical procedure that incises (opens) the armpit (axilla or axillary) to identify, examine, or remove lymph nodes (small glands, part of the lymphatic system, which filters cellular fluids).
Arm/Group | Vacuum Assisted Closure(Thigh) | Axillary Dissection(Thigh) | Vacuum Assisted Closure(Shank) | Axillary Dissection(Shank)
Number analyzed (Participants) | 36 | 36 | 36 | 36
participants | 1 | 4 | 15 | 5
Statistical Analysis 1: Comparison: Vacuum Assisted Closure(Thigh) vs Axillary Dissection(Thigh) vs Vacuum Assisted Closure(Shank) vs Axillary Dissection(Shank); Test type: Superiority or Other; p = 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Vacuum Assisted Closure(Thigh) | Axillary Dissection(Thigh) | Vacuum Assisted Closure(Shank) | Axillary Dissection(Shank)
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No